CLINICAL TRIAL: NCT00175487
Title: Femoral Head Resurfacing Versus a Large Femoral Head (Durom®) Total Hip System: A Prospective Randomized Trial
Brief Title: Comparison of Hip Resurfacing to Large Femoral Head Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H05-70105; C05-0105
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis; Avascular Necrosis
Keywords: Osteoarthritis/Avascular Necrosis; Hip
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Hip replacement — This study evaluates femoral head resurfacing versus a large femoral head (Durom®) total hip system. This is a prospective randomized trial.
  Other Names: Durom Total Hip System

SUMMARY:
This study evaluates femoral head resurfacing versus a large femoral head (Durom®) total hip system. This is a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for hip resurfacing because of osteoarthritis or avascular necrosis
2. Aged 19 to 65 years old
3. Ability to give informed consent

Exclusion Criteria:

1. Previous fracture requiring internal fixation of the hip
2. Previous hip osteotomy (pelvic or femoral)
3. Dysplasia requiring structural bone graft
4. Inability to respond to questionnaires in English (or French, Montreal centre only)
5. The presence of osteopenia or osteoporosis
6. Evidence of hepatic/renal insufficiency or failure from medical history or laboratory assessment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
To estimate the difference in postoperative quality of life between patients with Durom® hip resurfacing versus those with total hip arthroplasty (THA) using a large-head, metal-on-metal articulation | at 2 years

SECONDARY OUTCOMES:
To estimate the difference in concentrations of cobalt and chromium ions in serum
To estimate the difference in gait (pelvic tilt, forward velocity, and cadence) | at 12 and 52 weeks
To estimate the lower limb functional instability by a test of postural balance

CONTACTS AND LOCATIONS:
Overall Officials: Donald Garbuz, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada